CLINICAL TRIAL: NCT04073485
Title: Microwave Ablation for Uterine Fibroids
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor patient accrual
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-19-10
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave ablation (Other): The uterine fibroid will be identified and located with ultrasonography. A microwave electrode appropriate for the size of target lesion is placed into the target lesion under ultrasound guidance. Appropriate microwave power and application time are selected to provide sufficient ablation coverage to the target lesion.
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Microwave ablation — Ultrasonogram is performed to identify the fibroid or adenomyoma. A trocar needle is placed into the lesion under local anesthesia. The MWA procedure is performed using appropriate microwave power and application time are selected to provide sufficient ablation coverage to the target lesion.

SUMMARY:
This study is aimed to evaluate the clinical safety and effectiveness of Microwave ablation (MWA) in treating patients with uterine fibroid.

DETAILED DESCRIPTION:
Percutaneous radiofrequency ablation (RFA) is another form of thermal ablation that has been used for the treatment of uterine fibroids. Although RFA is more invasive when compared to High-Intensity-Focused-Ultrasound (HIFU), the treatment is less limited by the location of the lesions, and the treatment procedure is more time efficient. To further improve the technology of thermal ablation for uterine fibroid, percutaneous microwave ablation (MWA) could be a promising option because it allows increased efficiency of energy transmission and reduction in procedure time, and may allow effective treatment of large lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic fibroids with or without focal adenomyoma
2. Female gender
3. Age between 30 and 50
4. Pre or peri menopausal with FSH less than 40 mIU/ml
5. Negative urine pregnancy test
6. Uterine size less than 22 weeks based on physical exam assessment
7. Dominant intramural fibroid greater than or equal to 3 cm and less than or equal to 10 cm on imaging.
8. Good health other than history of leiomyomas. Chronic medications may be acceptable at the discretion of the research team.
9. Are using abstinence, mechanical (condoms, diaphragms) or sterilization methods of contraception and are willing to continue using them throughout the study.
10. Willing and able to give informed consent.
11. Willing and able to comply with study requirements.
12. Normal menstrual cycle with endometrial pathology excluded

Exclusion Criteria:

1. History of or current thromboembolic event (deep vein thrombosis, pulmonary embolus, stroke)
2. Other pelvic pathology as indicated by history or MR imaging such as endometriosis, ovarian tumor, acute or chronic pelvic inflammatory disease
3. Pregnant or Positive pregnancy test
4. Unexplained vaginal bleeding
5. Untreated severe cervical dysplasia
6. Abnormal adnexal /ovarian mass
7. Intrauterine device
8. Known recent rapid growth of fibroids, defined as a doubling in size in 6 months
9. Known bleeding tendency
10. Contraindication to MRI due to severe claustrophobia or implanted metallic device.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of technical success | within one hour
  Technical success was defined as successful completion of the planned treatment of target lesions

SECONDARY OUTCOMES:
Assessment of adverse effects and complications | up to 18 months
  Adverse effects and complications will be recorded during each treatment procedure, during each hospital admission related to the treatment, during each clinical visit at 1, 3, 6, 12 and 18 months
Assessment of volume change of the fibroids | 15 months after treatment
  Magnetic resonance imaging will be performed at 3 and 15 month after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Professor, Principal Investigator — DIIR, CUHK, Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No